CLINICAL TRIAL: NCT06830720
Title: A Non-interventional Study for Kisqali (Ribociclib) in Combination With an Aromatase Inhibitor for Adjuvant Treatment in Patients With HR+/HER2- Early Breast Cancer at High Risk of Recurrence to Evaluate Real-world Effectiveness, Safety Profile, Patient Compliance and Quality of Life
Brief Title: A Non-interventional Study for Kisqali (Ribociclib) in Combination With an Aromatase Inhibitor for Adjuvant Treatment in Patients With HR+/HER2- Early Breast Cancer at High Risk of Recurrence
Acronym: CAROLEEN
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011O1DE01
Record Dates: First submitted 2025-02-04; First posted 2025-02-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms
Keywords: Non-interventional study; NIS; breast cancer; early breast cancer; HR+; HER-; ribociclib; real world evidence; adjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; abemaciclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- ribociclib: ribociclib + AI ± LHRH
  Interventions: Drug: ribociclib + AI ± LHRH
- abemaciclib: abemaciclib + ET ± LHRH
  Interventions: Drug: abemaciclib + ET ± LHRH
- ET mono: ET mono ± LHRH
  Interventions: Drug: ET mono ± LHRH

INTERVENTIONS:
Drug: ribociclib + AI ± LHRH — ribociclib in combination with an aromatase inhibitor ± LHRH as described in the current effective summary of product characteristics. This is an observational study. There is no treatment allocation. The decision to initiate treatment will be based solely on clinical judgement.
  Groups: ribociclib
Drug: abemaciclib + ET ± LHRH — abemaciclib in combination with an endocrine therapy ± LHRH as described in the current effective summary of product characteristics. This is an observational study. There is no treatment allocation. The decision to initiate treatment will be based solely on clinical judgement.
  Groups: abemaciclib
Drug: ET mono ± LHRH — endocrine monotherapy ± LHRH. This is an observational study. There is no treatment allocation. The decision to initiate treatment will be based solely on clinical judgement.
  Groups: ET mono

SUMMARY:
This non-interventional observational study evaluates the real-world effectiveness and safety profile of ribociclib in combination with an aromatase inhibitor for adjuvant treatment in patients with HR+/HER2- early breast cancer at high risk of recurrence, as well as patient compliance and quality of life.

DETAILED DESCRIPTION:
This non-interventional study aims to provide information on real-world effectiveness, safety and tolerability, management of adverse events, QoL and patient compliance of patients with HR+/HER2- early breast cancer at high risk of recurrence treated with ribociclib in combination with an aromatase inhibitor (AI) ± luteinizing hormone-releasing hormone (LHRH) with curative intent according to the current effective local summary of product characteristics.

In order to put the results of patients treated with ribociclib into perspective, socio-economic data, data on QoL and patient compliance will also be collected from patients treated with abemaciclib + endocrine therapy (ET) ± LHRH as described in the current effective local summary of product characteristics.

To understand reasons for treatment decision, and to analyze the clinical adoption of ribociclib + AI ± LHRH after EU approval over time, baseline data will be collected from cohorts of ribociclib + AI ± LHRH, abemaciclib + ET ± LHRH, and additionally from patients treated with ET monotherapy ± LHRH and analyzed cross-sectionally.

The study is planned to be rolled out into a broad set of German and Austrian breast centers and gynecological practices to describe clinical routine in a representative subset of the local healthcare eco-system. It will gather insights into the potential benefits and risks associated with ribociclib + AI ± LHRH in the adjuvant treatment of HR+/HER2- eBC patients at high risk of recurrence. This knowledge will inform about clinical decision-making and contribute to improved patient outcomes in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of HR+/HER2- early breast cancer with curative intent
* Patients must have an indication for a treatment with ribociclib + AI ± LHRH as described in the current SmPC/"Fachinformation" of ribociclib (to be included into the cohorts of ribociclib + AI ± LHRH and ET mono ± LHRH) or abemaciclib + ET ± LHRH as described in the current SmPC/"Fachinformation" of abemaciclib (to be included into the abemaciclib + ET ± LHRH cohort) in the adjuvant setting
* Before enrollment the treating physician has made the decision in accordance with the patient to treat the patient with either

  * ribociclib + AI ± LHRH, or
  * ET mono ± LHRH, or
  * abemaciclib + ET ± LHRH and baseline is no longer than 2 weeks (14 days) prior to written informed consent for this study.

Baseline = for ribociclib + AI ± LHRH cohort: date of therapy start; for abemaciclib + ET ± LHRH cohort: date of therapy start; for ET mono ± LHRH cohort: within 4 weeks after therapy start or within 4 weeks after last non-endocrine based therapy, whichever is last.

* ≥18 years of age
* Written informed consent

Exclusion Criteria:

- Patient is simultaneously participating in any investigational trial or simultaneously participating in another Novartis-sponsored non-interventional study with ribociclib.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female and male patients with an indication for adjuvant treatment with ribociclib + AI ± LHRH (or abemaciclib + ET ± LHRH for the abemaciclib cohort) in HR+/HER2- eBC at high risk of recurrence as described in the current effective summary of product characteristics enrolled from specialized centers, hospitals and outpatient centers.
Sampling Method: Non-Probability Sample
Enrollment: 3250 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (iDFS) for adjuvant therapy with ribociclib + AI ± LHRH in participants with HR+/HER2- eBC at high risk of recurrence | 36 months
  iDFS using STEEP (Standardized Definitions for Efficacy Endpoints in Adjuvant Breast Cancer Trials) criteria, as assessed by the investigator. iDFS is defined as the time from study start to the date of the first event of invasive ipsilateral breast tumor recurrence, local/regional invasive recurrence, distant recurrence, death (any cause), contralateral invasive BC, or second primary non-breast invasive cancer (excluding basal and squamous cell carcinomas of the skin).

SECONDARY OUTCOMES:
Number of participants per Baseline parameters | baseline
  Description of available baseline characteristics (e.g. medical history, gender, menopausal status, disease characteristics, laboratory values, socio-economic status, genetic profile, etc.) by treatment cohorts
Reasons for treatment decision by treating physician | baseline
  Reason for treatment decision documented by the treating physician
Patients' individual perception of risk of recurrence and treatment decision | baseline
  Patients' individual perception of risk of recurrence and treatment decision assessed by questionnaire at baseline. The questionnaire is provided in two versions, with one version containing 6 items (applicable for the ET mono cohort), and the other version containing 11 items (applicable for ribociclib and abemaciclib cohorts). Responses are primarily given by selecting from predefined options, with some questions allowing multiple answers or prioritization. The scales and response options are designed to reflect individual preferences, concerns, and decision-making processes of patients. Higher scores on the importance scale indicate a stronger motivation to reduce recurrence risk
Invasive disease-free survival (iDFS) (ribociclib cohort) | 12 and 24 months
  iDFS using STEEP criteria. iDFS is defined as the time from study start to the date of the first event of invasive ipsilateral breast tumor recurrence, local/regional invasive recurrence, distant recurrence, death (any cause), contralateral invasive BC, or second primary non-breast invasive cancer (excluding basal and squamous cell carcinomas of the skin).
Invasive breast cancer-free survival (iBCFS) (ribociclib cohort) | 12, 24 and 36 months
  iBCFS using STEEP criteria. iBCFS is defined as the time from study start to the date of the first event of invasive ipsilateral breast tumor recurrence, local/regional invasive recurrence, distant recurrence, death (any cause), or contralateral invasive BC.
Recurrence-free survival (RFS) (ribociclib cohort) | 12, 24 and 36 months
  RFS using STEEP criteria. RFS is defined as the time from study start to the date of the first event of invasive ipsilateral breast tumor recurrence, local/regional invasive recurrence, distant recurrence, or death (any cause).
Distant disease-free survival (DDFS) (ribociclib cohort) | 12, 24 and 36 months
  DDFS using STEEP criteria. DDFS is defined as the time from study start to the date of the first event of distant recurrence, death (any cause), or second primary non-breast invasive cancer (excluding basal and squamous cell carcinomas of the skin).
Incidence and severity of adverse events (ribociclib cohort) | up to 36 months
  Incidence and severity of adverse events
Dose modification rates (ribociclib cohort) | up to 36 months
  Proportion of patients with dose modification and underlying cause
Treatment interruption rates (ribociclib cohort) | up to 36 months
  Proportion of patients with treatment interruption and underlying cause
Discontinuation rates (ribociclib cohort) | up to 36 months
  Proportion of patients who discontinued treatment and underlying cause
Time to discontinuation (TTD) (ribociclib cohort) | up to 36 months
  Time from treatment start to permanent treatment discontinuation
Quality of life by EORTC QLQ-C30 (ribociclib and abemaciclib cohorts) | up to 39 months
  Changes from baseline as assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30. The EORTC QLQ-C30 is a participant completed 30 item questionnaire that is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, six single items and a GHS/QoL scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life by EORTC QLQ-BR42 (ribociclib and abemaciclib cohorts) | up to 39 months
  Changes from baseline as assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-BR42. The Breast Cancer Module EORTC QLQ-BR42 is a 42 item instrument designed to measure quality of life in breast cancer participants. It includes three functional scales, six symptom scales and three single items. All the scales and single item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life by HADS D (ribociclib and abemaciclib cohorts) | up to 39 months
  Changes from baseline as assessed by the Hospital Anxiety and Depression Scale (HADS D). The HADS is a participant completed fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains.
Participant compliance as assessed by the Medication Adherence Report Scale (MARS-D) (ribociclib and abemaciclib cohorts) | up to 36 months
  Medication Adherence Report Scale (MARS-D) questionnaire is a 5-item questionnaire measuring non-adherence. Each item is ranging from "never" (5 points) to "always" (1 point), with a total score 5-25 where higher scores indicate better compliance.
Participant compliance as assessed by a physician adherence rating (ribociclib cohort) | up to 36 months
  Participant compliance as assessed by a physician adherence rated as very good, good, moderate, or poor.
Participant compliance as assessed by neutrophil count (ribociclib cohort) | up to 36 months
  Participant compliance as assessed by neutrophil count.
Impact of type and change of treatment facility and health care professionals involved in treatment management on participant compliance assessed by MARS-D (ribociclib cohort) | up to 36 months
  Medication Adherence Report Scale (MARS-D) questionnaire is a 5-item questionnaire measuring non-adherence. Each item is ranging from "never" (5 points) to "always" (1 point), with a total score 5-25 where higher scores indicate better compliance.
Impact of digital health solutions applied in clinical routine on participant compliance assessed by MARS-D (ribociclib cohort) | up to 36 months
  Medication Adherence Report Scale (MARS-D) questionnaire is a 5-item questionnaire measuring non-adherence. Each item is ranging from "never" (5 points) to "always" (1 point), with a total score 5-25 where higher scores indicate better compliance.
Socio-economic status of participants measured by WPAI-GH (ribociclib and abemaciclib cohorts) | up to 39 months
  The Work Productivity and Activity Impairment - General Health questionnaire (WPAI-GH) is a participant completed 6 item questionnaire which addresses absenteeism, presenteeism, overall work productivity loss, and activity impairment for the 7 days prior to the assessment. WPAI outcomes are presented as impairment percentages (range goes from 0 to 100 with a higher percentage indicating greater impairment and less productivity).
Number of participants per reason for treatment discontinuation (ribociclib and abemaciclib cohorts) | up to 39 months
  Reported reasons for treatment discontinuation
Type of subsequent anti-neoplastic therapies (ribociclib and abemaciclib cohorts) | up to 39 months
  Type of subsequent anti-neoplastic therapies will be recorded
Time to subsequent anti-neoplastic therapy (ribociclib and abemaciclib cohorts) | up to 39 months
  Time from study start to first subsequent anti-neoplastic therapy
Impact of an active participation of the participant in the treatment decision on subsequent participant compliance measured by MARS-D (ribociclib cohort) | up to 36 months
  Participant compliance assessed by MARS-D and active participation of the participant in the treatment decision assessed by the questionnaire "Fragebogen zur partizipativen Entscheidungsfindung aus Participantensicht" (PEF-FB-9) and "Fragebogen zur partizipativen Entscheidungsfindung aus Sicht des Arztes"(PEF-FB-Doc) at baseline.
  The MARS-D is a 5-item questionnaire measuring non-adherence with a total score of 5-25 where higher scores indicate better compliance.
  The PEF-FB-9 is a participant completed 9 item questionnaire for participant participation in decision-making. The 9 items are rated on a 6-point scale with endpoints ranging from "does not apply at all" to "applies completely", summed up and transformed into a scale from 0 to 100. The higher the total score, the higher the perceived degree of participation.
  The PEF-FB-Doc is the physician version of the PEF-FB-9.
  The correlation between participation on treatment decisions and participant compliance will be presented.
Impact of participants' fear of cancer recurrence on participant compliance measured by MARS-D (ribociclib cohort) | up to 36 months
  Participant compliance assessed by MARS-D and participants' fear of cancer recurrence assessed by the Fear of Cancer Recurrence (FCR)-1 questionnaire.
  The MARS-D questionnaire is a 5-item questionnaire measuring non-adherence. Each item is ranging from "never" (5 points) to "always" (1 point), with a total score 5-25 where higher scores indicate better compliance.
  The FCR-1 is a participant completed 1 item questionnaire asking the participant to describe their subjective level of fear of cancer recurrence at the given time on a scale from 0 to 100 with 100 being the greatest fear.
  The correlation between participants' fear of recurrence and participant compliance will be presented.
Participants' expectations regarding therapy, side effects and management (ribociclib and abemaciclib cohorts) | baseline
  Treatment expectation assessed by a questionnaire containing 5 questions with each 5-7 ordinal answer categories with the same directionality on participants' expectations regarding therapy, side effects and management
Participants' treatment satisfaction (ribociclib and abemaciclib cohorts) | up to 24 months
  Treatment satisfaction assessed by a questionnaire containing 5 questions with each 5-7 ordinal answer categories with the same directionality on treatment satisfaction

CONTACTS AND LOCATIONS:
Locations (223):
- Austria (8):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Linz, Upper Austria
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Klagenfurt
  - Novartis Investigative Site, Leoben
  - Novartis Investigative Site, Schwaz
  - Novartis Investigative Site, Steyr
  - Novartis Investigative Site, Vienna
- Germany (215):
  - Novartis Investigative Site, Filderstadt, Baden-Wurttemberg
  - Novartis Investigative Site, Freudenstadt, Baden-Wurttemberg
  - Novartis Investigative Site, Heidenheim, Baden-Wurttemberg
  - Novartis Investigative Site, Konstanz, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Nürtingen, Baden-Wurttemberg
  - Novartis Investigative Site, Ostfildern, Baden-Wurttemberg
  - Novartis Investigative Site, Pforzheim, Baden-Wurttemberg
  - Novartis Investigative Site, Ravensburg, Baden-Wurttemberg
  - Novartis Investigative Site, Reutlingen, Baden-Wurttemberg
  - Novartis Investigative Site, Schwaebisch, Baden-Wurttemberg
  - Novartis Investigative Site, Winnenden, Baden-Wurttemberg
  - Novartis Investigative Site, Altötting, Bavaria
  - Novartis Investigative Site, Ansbach, Bavaria
  - Novartis Investigative Site, Augsburg, Bavaria
  - Novartis Investigative Site, Bayreuth, Bavaria
  - Novartis Investigative Site, Donauwörth, Bavaria
  - Novartis Investigative Site, Ebersberg, Bavaria
  - Novartis Investigative Site, Erlangen, Bavaria
  - Novartis Investigative Site, Fürth, Bavaria
  - Novartis Investigative Site, Herrsching am Ammersee, Bavaria
  - Novartis Investigative Site, Kempten (Allgäu), Bavaria
  - Novartis Investigative Site, Kronach, Bavaria
  - Novartis Investigative Site, Landsberg am Lech, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Rosenheim, Bavaria
  - Novartis Investigative Site, Traunstein, Bavaria
  - Novartis Investigative Site, Waldmuenchen, Bavaria
  - Novartis Investigative Site, Weilheim, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Brandenburg, Brandenburg
  - Novartis Investigative Site, Cottbus, Brandenburg
  - Novartis Investigative Site, Königs Wusterhausen, Brandenburg
  - Novartis Investigative Site, Bremen, City state Bremen
  - Novartis Investigative Site, Bremerhaven, City state Bremen
  - Novartis Investigative Site, Schwerte, Germany
  - Novartis Investigative Site, Hamburg, Hamburg
  - Novartis Investigative Site, Bad Homburg, Hesse
  - Novartis Investigative Site, Bad Nauheim, Hesse
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Langen, Hesse
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Wiesbaden, Hesse
  - Novartis Investigative Site, Braunschweig, Lower Saxony
  - Novartis Investigative Site, Georgsmarienhütte, Lower Saxony
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Hildesheim, Lower Saxony
  - Novartis Investigative Site, Ilsede, Lower Saxony
  - Novartis Investigative Site, Lingen Ems, Lower Saxony
  - Novartis Investigative Site, Osnabrück, Lower Saxony
  - Novartis Investigative Site, Twistringen, Lower Saxony
  - Novartis Investigative Site, Westerstede, Lower Saxony
  - Novartis Investigative Site, Wolfenbüttel, Lower Saxony
  - Novartis Investigative Site, Wunstorf, Lower Saxony
  - Novartis Investigative Site, Rostock, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Bergisch Gladbach, North Rhine-Westphalia
  - Novartis Investigative Site, Bielefeld, North Rhine-Westphalia
  - Novartis Investigative Site, Bochum, North Rhine-Westphalia
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Dortmund, North Rhine-Westphalia
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Mönchengladbach, North Rhine-Westphalia
  - Novartis Investigative Site, Olpe, North Rhine-Westphalia
  - Novartis Investigative Site, Paderborn, North Rhine-Westphalia
  - Novartis Investigative Site, Remscheid, North Rhine-Westphalia
  - Novartis Investigative Site, Siegen, North Rhine-Westphalia
  - Novartis Investigative Site, Troisdorf, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Remscheid Innen, Northrhine Westfalia
  - Novartis Investigative Site, Speyer, Rhineland-Palatinate
  - Novartis Investigative Site, Lebach, Saarland
  - Novartis Investigative Site, Borna, Saxony
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Neustadt in Sachsen, Saxony
  - Novartis Investigative Site, Radebeul, Saxony
  - Novartis Investigative Site, Rodewisch, Saxony
  - Novartis Investigative Site, Salzwedel, Saxony
  - Novartis Investigative Site, Scheibenberg, Saxony
  - Novartis Investigative Site, Schkeuditz, Saxony
  - Novartis Investigative Site, Zittau, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Magdeburg, Saxony-Anhalt
  - Novartis Investigative Site, Stendal, Saxony-Anhalt
  - Novartis Investigative Site, Flensburg, Schleswig-Holstein
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Berlin, State of Berlin
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Mühlhausen, Thuringia
  - Novartis Investigative Site, Nordhausen, Thuringia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Amberg
  - Novartis Investigative Site, Apolda
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Friedrichshall
  - Novartis Investigative Site, Bad Langensalza
  - Novartis Investigative Site, Bad Mergentheim
  - Novartis Investigative Site, Bad Reichenhall
  - Novartis Investigative Site, Bad Soden
  - Novartis Investigative Site, Baden-Baden
  - Novartis Investigative Site, Balingen
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Bautzen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Biberach
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Brandenburg
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Bremerhaven
  - Novartis Investigative Site, Bruchsal
  - Novartis Investigative Site, Celle
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Coburg
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dachau
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dillingen A D Donau
  - Novartis Investigative Site, Dorfen
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eggenfelden
  - Novartis Investigative Site, Ehingen
  - Novartis Investigative Site, Ehrenfriedersdorf
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Eschweiler
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Fürstenwalde
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Gerlingen
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Gummersbach
  - Novartis Investigative Site, Günzburg
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Haldensleben I
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heide
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Hennigsdorf
  - Novartis Investigative Site, Herdecke
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Krefeld
  - Novartis Investigative Site, Kulmbach
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Loerrach
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marktredwitz
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Moers
  - Novartis Investigative Site, Mutlangen
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Naunhof
  - Novartis Investigative Site, Neubrandenburg
  - Novartis Investigative Site, Neuss
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Offenburg
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Passau
  - Novartis Investigative Site, Plauen Kauschwitz
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Prien A Chiemsee
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Rendsburg
  - Novartis Investigative Site, Rheine
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rotenburg (Wümme)
  - Novartis Investigative Site, Rüsselsheim am Main
  - Novartis Investigative Site, Saalfeld
  - Novartis Investigative Site, Saarlouis
  - Novartis Investigative Site, Schorndorf
  - Novartis Investigative Site, Schweinfurt
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Sigmaringen
  - Novartis Investigative Site, Singen
  - Novartis Investigative Site, Sinsheim
  - Novartis Investigative Site, Soest
  - Novartis Investigative Site, Stendal
  - Novartis Investigative Site, Stralsund
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Suhl
  - Novartis Investigative Site, Torgau
  - Novartis Investigative Site, Traunstein
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Villingen
  - Novartis Investigative Site, Waldkirchen
  - Novartis Investigative Site, Waldsassen
  - Novartis Investigative Site, Walsrode
  - Novartis Investigative Site, Weiden
  - Novartis Investigative Site, Weinheim
  - Novartis Investigative Site, Werdau
  - Novartis Investigative Site, Wernigerode
  - Novartis Investigative Site, Wesel
  - Novartis Investigative Site, Wetzlar
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Winse Luhe
  - Novartis Investigative Site, Witten
  - Novartis Investigative Site, Worms
  - Novartis Investigative Site, Würzburg